CLINICAL TRIAL: NCT02036099
Title: Driving in Mild Dementia Decision Tool
Acronym: DMD-DT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAL129896
Record Dates: First submitted 2014-01-03; First posted 2014-01-14 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Dementia
Keywords: Dementia; Automobile driving; Accidents, traffic
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will assess patients using the Driving in Mild Dementia Decision Tool.
  Interventions: Other: Driving in Mild Dementia Decision Tool
- Control (No Intervention): Participants in this arm will assess patients using their usual care strategies.

INTERVENTIONS:
Other: Driving in Mild Dementia Decision Tool
  Arms: Intervention

SUMMARY:
Based on the literature on dementia and driving, and on knowledge tools available to date including one from our current work, a Driving in Mild Dementia Decision Tool (DMD-DT) will be adapted and tailored to guide physicians in their decisions to report a driver with mild dementia to the provincial licensing agency. The DMD-DT intervention will include a) an algorithm-based computerized clinical decision support system (CCDSS) for facilitating driving assessment and physicians' reporting to provincial transportation authorities, b) an individualized educational package for patients and caregivers about dementia and driving and driving cessation, and c) a modified reporting form to provincial driving regulatory authorities. Months 1 to 6: The DMD-DT will be tailored and adapted to practice with the input of the co-investigators and knowledge-users who represent the perspectives of physicians, patients and their caregivers, as well as transportation authorities. Pilot testing will be done, and input from focus groups of knowledge-users will refine the intervention. Physicians will be recruited to participate in a clinical trial of the DMD-DT. Months 7-18: A parallel-group cluster randomized controlled trial (RCT) will be conducted to compare the effects of the DMD-DT to a legislation reminder on recommendations for reporting to the licensing agency. The effects of the DMD-DT on the doctor-patient relationship will be further explored in focus groups and interviews with physicians. Months 19-24: The knowledge obtained from the study will be used to generalize and sustain use of the intervention beyond Ontario, Canada, and to disseminate the information to knowledge-users. The primary outcome measure is the filing of a report to the Ministry of Transportation of Ontario, indicating that the physician has a concern about the patient's health condition (i.e. mild dementia). The primary outcome of the study is the difference in reporting between the DMD-DT and control arms. Since the current reporting rate is low, approximately 13%, from a public health point of view, the primary outcome expected is that physicians in the DMD-DT group will report more patients with mild dementia than those in the control group.

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* family physicians and specialist physicians (geriatricians, geriatric psychiatrists, cognitive neurologists) practicing in Ontario, Canada, who assess and treat patients with mild dementia
* must speak English and have computer access at the point of delivery of care

Exclusion Criteria:

* family physicians must see at least 10 new patients per year with mild dementia, and specialist physicians must see at least 12 new patients per year with mild dementia
* participants must not have participated in, attended a continuing medical education (CME) event about, or read about our "Dementia and Driving in Ontario" study (2010-2012)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients reported to the Ontario Ministry of Transportation | When participants have completed 500 patient assessments (expected to take approximately 12 months)
  The primary outcome of this study is the number of patients reported to the Ontario Ministry of Transportation by study participants. A "report" indicates that the participant believes his/her patient may be unsafe to continue driving due to mild cognitive impairment or mild dementia. The difference in the number of reports filed between the intervention and control group participants will be assessed.

SECONDARY OUTCOMES:
The number of "false positives", i.e. number of patients reported to the Ontario Ministry of Transportation as potentially being unsafe drivers who are deemed by expert consensus to be safe drivers. | When participants have completed 500 patient assessments (expected to take approximately 12 months)
  Although the primary aim of the study from a public health point of view is to increase reporting of patients with mild dementia to transportation authorities who are unsafe to drive according to best-evidence, it is important to ensure that physician reporting does not unfairly punish those who are deemed not to be at significant potential risk. Hence, a secondary outcome measure will examine the number of false positive reports, or the number of patients reported when expert consensus indicates they should NOT be reported.
Number of recommendations given for specialized on-road testing | When participants have completed 500 patient assessments (expected to take approximately 12 months)
  International guidelines suggest that when physicians are uncertain about the driving safety of their patients, specialized on-road testing should be strongly considered. Such testing, while expensive, has substantially more face validity than in-office testing. A secondary outcome measure for this study is therefore the number of recommendations made by participants for specialized on-road testing for the patients assessed in the study.
Quality of Doctor-Patient Relationship | When participants have completed 500 patient assessments (expected to take approximately 12 months)
  Many physicians avoid discussing issues related to driving with their patients who have mild dementia and their caregivers or family members, because it can have a negative effect on the doctor-patient relationship. The impact of the Driving in Mild Dementia Decision Tool on the doctor-patient relationship will be examined in two ways: first, by comparing responses between intervention and control group participants on four 5-point Likert-type questions following each patient encounter; and second, by analyzing transcripts from focus groups with participants following completion of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Rapoport, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rapoport MJ, Zucchero Sarracini C, Kiss A, Lee L, Byszewski A, Seitz DP, Vrkljan B, Molnar F, Herrmann N, Tang-Wai DF, Frank C, Henry B, Pimlott N, Masellis M, Naglie G. Computer-Based Driving in Dementia Decision Tool With Mail Support: Cluster Randomized Controlled Trial. J Med Internet Res. 2018 May 25;20(5):e194. doi: 10.2196/jmir.9126. PMID 29802093